CLINICAL TRIAL: NCT04235790
Title: Examining Behaviors of Teachers of Invasive Bedside Procedures Using an Eye Tracking Device: Towards Improving Supervisor Expertise and Decreasing Complications in the Intensive Care Unit
Brief Title: Examining Behaviors of Teachers of Invasive Bedside Procedures Using an Eye Tracking Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Diana J. Kelm, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-003774
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Procedural Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Student or Resident (No Intervention): Subjects will perform simulated central venous catheters (CVC) insertions.
- Novice and Expert IBP Teachers (Other): Expert teachers will be identified based on years as faculty, number of supervised procedures, prior teacher awards, and participation in IBP teaching at international conferences. Novice teachers will include those that have performed less than 50 CVCs. Teachers will supervise 3 simulated central venous catheters (CVC) insertions with increased complexity while wearing an eye tracking device.
  Interventions: Device: Eye Tracking Device

INTERVENTIONS:
Device: Eye Tracking Device — Eye tracking glasses
  Other Names: Tobii Pro Glasses 2.0
  Arms: Novice and Expert IBP Teachers

SUMMARY:
Researchers are studying the behaviors in teachers of invasive bedside procedures to improve the safety of invasive bedside procedure in the Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Novice and expert Invasive bedside procedure (IBP) teachers from Pulmonary Critical Care Medicine and Anesthesia-Critical Care at Mayo Clinic Rochester
* Expert teachers will be identified based on years as faculty, number of supervised procedures, prior teacher awards, and participation in IBP teaching at international conferences
* Novice teachers will include those that have performed less than 50 CVCs
* Medical student or resident

Exclusion Criteria:

* <25% FTE in the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Fixation Frequency | Duration of procedure (approximately 4 hours)
  Number of fixations within an area of interest. Higher values indicate focused attention.
Visit Frequency | Duration of procedure (approximately 4 hours)
  Number of times an area of interest is entered and left. Indexes which areas repeatedly attracted participant's attention.
Dwell Time | Duration of procedure (approximately 4 hours)
  Total fixation duration measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Diana Kelm, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials